CLINICAL TRIAL: NCT00835172
Title: A Relative Bioavailability Study of Glimepiride 4 mg Tablets Under Non-Fasting Conditions
Brief Title: Glimepiride 4 mg Tablets Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B036502
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glimepiride (Experimental): Glimepiride 4 mg Tablet (test) dosed in first period followed by Amaryl® 4 mg Tablet (reference) dosed in second period
  Interventions: Drug: Glimepiride 4 mg Tablets
- Amaryl® (Active Comparator): Amaryl® 4 mg Tablet (reference) dosed in first period followed by Glimepiride 4 mg Tablet (test) dosed in second period
  Interventions: Drug: AMARYL® 4 mg Tablets

INTERVENTIONS:
Drug: Glimepiride 4 mg Tablets — 1 x 4 mg, single-dose non-fasting
  Arms: Glimepiride
Drug: AMARYL® 4 mg Tablets — 1 x 4 mg, single-dose non-fasting
  Arms: Amaryl®

SUMMARY:
The objective of this study is to compare the relative bioavailability of glimepiride 4 mg tablets (manufactured by TEVA Pharmaceutical Industries, Ltd. and distributed by TEVA Pharmaceuticals USA) with that of AMARYL® tablets (Aventis) in healthy, adult, non-smoking subjects under non-fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* All subjects selected for this study will be non-smokers at least 18 years of age. Subjects will have a BMI (body mass index) of 30 or less.
* Each subject shall be given a general physical examination within 28 days of initiation of the study. Such examination includes, but is not limited to, blood pressure, general observations, and history.
* Each female subject will be given a serum pregnancy test as part of the pre-study screening process.

Adequate blood and urine samples should be obtained within 28 days before beginning of the first period and at the end of the trial for clinical laboratory measurements.

Clinical laboratory measurements will include the following:

* Hematology: hemoglobin, hematocrit, red blood cell count, platelets, whit blood cell count (with differential).
* Clinical Chemistry: creatinine, BUN, glucose, SGOT/AST, SGPT/ALT, bilirubin, and alkaline phosphatase.
* Urine Analysis: pH, specific gravity, protein, glucose, ketones, bilirubin, occult blood, and cells.
* HIV Screen: pre-study only.
* Hepatitis-B, C Screen: pre-study only.
* Drugs of Abuse Screen: pre-study and at each check-in. Subjects will be selected if all above are normal.

Exclusion Criteria:

* Subjects with a significant recent history of chronic alcohol consumption, drug addiction, or serious gastrointestinal, renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma, diabetes, psychosis or glaucoma will not be eligible for this study.
* Subjects whose clinical laboratory test values are greater than 20% outside the normal range may be retested. If the clinical values are outside the range on retesting, the subject will not be eligible to participate in the study unless the clinical investigator deems the result to not be significant.
* Subjects who have a history of allergic responses to the class of drug being tested will be excluded from the study.
* Subjects who use tobacco in any form will not be eligible to participate in the study. Three months abstinence is required.
* All subjects will have urine samples assayed for the presence of drugs of abuse as part of the clinical laboratory screening procedures and at each dosing period check-in. Subjects found to have urine concentrations of any of the tested drugs will not be allowed to participate.
* Subjects should not have donated blood and/or plasma for at least thirty (30) days prior to the first dosing of the study.
* Subjects who have taken any investigational drug within thirty (30) days prior to the first dosing of the study will not be allowed to participate.
* Female subjects who are pregnant, breast-feeding, or who are likely to become pregnant during the study will not be allowed to participate. Female subjects of childbearing potential must either abstain from sexual intercourse or use a reliable barrier method (e.g. condom, IUD) of contraception during the course of the study (first dosing until last blood collection) or they will not be allowed to participate. Female subjects who have used hormonal oral contraceptives within 14 days of dosing or implanted or injected hormonal contraceptives within 180 days of dosing will not be allowed to participate.
* All female subjects will be screened for pregnancy at check-in each study period. Subjects with positive or inconclusive results will be withdrawn from the study.
* Subjects who do not tolerate venipuncture will not be allowed to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2003-03; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Solomon G. Ghide, M.D., Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceutical Research Services, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Glimepiride (Test) First: Glimepiride 4 mg Tablet (test) dosed in first period followed by Amaryl® 4 mg Tablet (reference) dosed in second period
- Amaryl® (Reference) First: Amaryl® 4 mg Tablet (reference) dosed in first period followed by Glimepiride 4 mg Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Glimepiride (Test) First | Amaryl® (Reference) First
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Washout
Arm/Group | Glimepiride (Test) First | Amaryl® (Reference) First
Started | 16 | 16
Completed | 16 | 15
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Second Intervention
Arm/Group | Glimepiride (Test) First | Amaryl® (Reference) First
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glimepiride (Test) First | Amaryl® (Reference) First | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 10 | 6 | 16
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 6 | 3 | 9
  Black | 8 | 9 | 17
  Hispanic | 2 | 3 | 5
  Biracial | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Glimepiride: Glimepiride 4 mg Tablet (test) dosed in either period
- Amaryl®: Amaryl® 4 mg Tablet (reference) dosed in either period
Arm/Group | Glimepiride | Amaryl®
Number analyzed (Participants) | 31 | 31
ng/mL | 267.629 (101.151) | 266.706 (107.927)
Statistical Analysis 1: Comparison: Glimepiride vs Amaryl®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Geometric Test/Ref Ratio x 100 = 102, 90% CI [92.1 to 112] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUCinf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUCinf
Time Frame: Blood samples collected over 24 hour period
Population: The parameter of AUCinf could not be estimated for three subjects.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Glimepiride | Amaryl®
Number analyzed (Participants) | 28 | 28
ng*h/mL | 1751.420 (1071.151) | 1824.742 (1346.454)
Statistical Analysis 1: Comparison: Glimepiride vs Amaryl®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Geometric Test/Ref Ratio x 100 = 101, 90% CI [96.8 to 105] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Glimepiride | Amaryl®
Number analyzed (Participants) | 31 | 31
ng*h/mL | 1639.083 (846.547) | 1632.301 (969.908)
Statistical Analysis 1: Comparison: Glimepiride vs Amaryl®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Geometric Test/Ref Ratio x 100 = 103, 90% CI [99.3 to 106] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.